CLINICAL TRIAL: NCT05834660
Title: SAFETY-A for Promoting Equity in Suicide Prevention Outcomes in Schools
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Anna Lau, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 092530369
Record Dates: First submitted 2023-04-13; First posted 2023-04-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: Suicidal Ideation
Keywords: Implementation Feasibility; Implementation Acceptability
MeSH Terms: conditions — Suicidal Ideation | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safe Alternatives for Teens and Youth-Acute for Schools (SAFETY-A for Schools) (Experimental): SAFETY-A is a brief, family centered, cognitive-behavioral approach to therapeutic risk assessment and safety planning that can be delivered via school-based providers. The intervention is delivered in one session during which the youth at risk for suicidal behavior works with the provider to identify strengths, supports, understand emotional antecedents and warning signs, identify alternative coping behaviors and thoughts, and ways to keep the environment safe. Youth and families receive follow-up contacts after the SAFETY-A session. The primary focus is on the therapeutic mechanisms of hope, reduced intensity of suicidal urges, increased confidence in ability to keep safe. Adaptation of SAFETY-A for Schools will target mechanisms that are presumed to drive disparities in mental health service use among Asian American and Latinx youth: (1) trust in mental health services, (2) internalized stigma, and (3) comfort communicating distress.
  Interventions: Behavioral: Safe Alternatives for Teens and Youth-Acute for Schools (SAFETY-A for Schools)

INTERVENTIONS:
Behavioral: Safe Alternatives for Teens and Youth-Acute for Schools (SAFETY-A for Schools) — SAFETY-A is a brief, family centered, cognitive-behavioral approach to therapeutic risk assessment and safety planning that can be delivered via school-based providers. The intervention is delivered in one session during which the youth at risk for suicidal behavior works with the provider to identify strengths, supports, understand emotional antecedents and warning signs, identify alternative coping behaviors and thoughts, and ways to keep the environment safe. Youth and families receive follow-up contacts by phone at 1, 2, and 4 weeks after the SAFETY-A session. The primary focus is on the therapeutic mechanisms of hope, reduced intensity of suicidal urges, increased confidence in ability to keep safe. Adaptation of SAFETY-A for Schools will target mechanisms that are presumed to drive disparities in mental health service use among Asian American and Latinx youth: (1) trust in mental health services, (2) internalized stigma, and (3) comfort communicating distress.

SUMMARY:
This study will adapt Safe Alternatives For Teens and Youth - Acute (SAFETY-A) for implementation in low-resourced school districts to reduce racial/ethnic disparities in mental health service use (MHS) following identification of suicide risk in youth. SAFETY-A will be adapted to fit the organizational context of school districts and to reduce mistrust of MHS, internalized stigma, and concealment of youth emotional distress that arise in school suicide risk assessments with Asian American and Latinx students. Following a prototyping case series, a feasibility trial will assign four districts to the timing of SAFETY-A implementation to generate preliminary data on feasibility and impacts on proposed mechanisms and youth MHS utilization and clinical outcomes across racial/ethnic groups.

DETAILED DESCRIPTION:
The proposed study will adapt Safe Alternatives For Teens and Youth - Acute (SAFETY-A) for implementation in low-resourced school districts to target putative mechanisms underlying disparities in MHS use following youth suicide risk detection. SAFETY-A will be adapted to reduce mistrust of MHS, internalized stigma, and concealment of youth emotional distress that drive poor engagement in MHS among Asian American and Latinx students and families. Furthermore, SAFETY-A delivery parameters and implementation strategies will be adapted to fit the organizational context of school district policies and protocols, resource constraints, and workforce needs.

The proposed intervention development study will include three phases. First, stakeholders will be engaged to design adaptations to the intervention and implementation strategy. Provider, youth and caregiver input will be gathered using human-centered design approaches to adapting the SAFETY-A intervention content to address disparities mechanisms. School district leaders, school administrators, and MHS providers will help to develop a tailored implementation strategy to fit local training and support needs across a range of district contexts. Second, a prototyping case series will inform iterative refinements of SAFETY-A in one school district. Third, a pilot feasibility trial will assign school districts to the timing of implementation to provide preliminary data on the implementation outcomes of provider adherence, and perceptions of feasibility, acceptability and fit. The proposed project will provide preliminary data on feasibility and potential impacts on putative mechanisms to propose a definitive Hybrid Type 1 trial to test SAFETY-A as an intervention to reduce racial/ethnic disparities in MHS utilization among suicidal youth.

ELIGIBILITY:
Inclusion Criteria:

1. Age 11-19
2. Enrolled in participating school district
3. Present with suicide thoughts or behavior to school personnel
4. Have an identified caregiver who can participate in the intervention

Exclusion Criteria:

1. School personnel determine the student to be at such imminent risk of danger to self that they are unable to benefit from the intervention and must be immediate transported for emergency care.
2. Student is unable to participate in the intervention due to indications of intellectual disability, psychosis, or intoxication

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Referral Tracking System (Kim et al., 2018) | Six months following the intervention
  As described in Kim, Kodish, Bear, El-Hendi, Duong & Lau (2018), we will extract mental health service use outcomes from administrative records maintained by each school district. The variable of interest will be Linkage to Outpatient Care, indexed by a receipt of at least one outpatient session following referral to care.

SECONDARY OUTCOMES:
SAFE Alternatives for Teens and Youths - Acute Pre-to-Post intervention Questionnaire (Zullo et al., 2020). | Change in youth ratings from beginning of the intervention session to the end of the intervention session.
  As described in Zullo, Meza, Rolon-Aroyoo, Vargas, Venables, Miranda & Asarnow (2020). Youths are asked to rate the intensity of their suicide urge, feelings of hope, and ability to keep safe on a scale from 1-5 at the beginning and end of session.

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Lau, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified individual level data will be shared according to the National Data Archive data submission plan.